CLINICAL TRIAL: NCT07011849
Title: A Multi-center, Open-label Phase II Study of Lenvatinib Plus Pembrolizumab (LEAP) in Renal Cell Carcinoma Patients With Brain Metastasis Previously Treated With Immune Checkpoint Blockade
Brief Title: Study of Lenvatinib Plus Pembrolizumab in IO Refractory mRCC Patients With Brain Metastases
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: 0 participants
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0331; NCI-2025-04029 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Renal Cell Carcinoma; Brain Metastasis
MeSH Terms: conditions — Carcinoma, Renal Cell; Brain Neoplasms | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Second Course: Retreatment with Pembrolizumab (Experimental)
  Interventions: Drug: Pembrolizumab
- Treatment with Pembrolizumab and Lenvatinib (Experimental)
  Interventions: Drug: Pembrolizumab; Drug: Lenvatinib

INTERVENTIONS:
Drug: Pembrolizumab — Given by IV
Drug: Lenvatinib — Given by mouth
  Arms: Treatment with Pembrolizumab and Lenvatinib

SUMMARY:
This is a multi-center, open-label phase II study evaluating the efficacy and safety of pembrolizumab in combination with lenvatinib in patients with renal cell carcinoma (RCC) and brain metastasis who were previously treated with immune checkpoint blockade.

DETAILED DESCRIPTION:
Primary Objectives:

Primary Objective: To determine the intracranial PFS of pembrolizumab plus lenvatinib in IO refractory mRCC participants with brain metastases per Response Assessment in Neuro-Oncology-Brain Metastases (RANO-BM) criteria (Appendix 1).

Hypothesis: Investigators hypothesize that pembrolizumab plus lenvatinib will provide a higher intracranial PFS in RCC participants with brain metastases when compared to historical data.

Primary Endpoint: intracranial PFS per RANO-BM criteria.

Secondary Objectives:

* To determine the intracranial ORR in participants with remaining non-irradiated brain metastases, as assessed by RANO-BM criteria.
* To determine the local control rate in participants with irradiated brain metastases at 1 year, as assessed by RANO-BM criteria.
* To determine the rate of new brain metastasis at a site different from the original brain metastases at 1 year (Distant brain failure rate), as assessed by RANO-BM criteria.
* To determine the intracranial disease control rate: complete response + partial response + stable disease (DCR: CR + PR + SD) in participants with remaining non-irradiated brain metastases, as assessed by RANO-BM.
* To determine the intracranial clinical benefit rate (CBR: CR + PR + .6 months SD) in participants with remaining non-irradiated brain metastases, as assessed by RANO-BM.
* To determine the intracranial duration of response (DOR) in participants with remaining nonirradiated brain metastases, as assessed by the RANO-BM.
* To determine the time to response (TTR) in participants with remaining non-irradiated brain metastases, as assessed by the RANO-BM.
* To evaluate the safety and tolerability, as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 (Appendix 9).
* To define symptomatic radiation necrosis rate defined as the rate of clinical symptomatology requiring steroid administration and/or operative intervention concomitant with advanced and routine brain imaging findings consistent with radiation necrosis.
* To determine the extracranial ORR, as assessed by the Modified Response Evaluation Criteria in Solid Tumors v1.1 (RECIST 1.1).
* To determine extracranial PFS, as assessed by the RECIST 1.1 and iRECIST.
* To determine bi-compartmental PFS, as assessed by RECIST 1.1 and iRECIST for extracranial disease and RANO-BM for intracranial disease.
* To evaluate OS.

Secondary Endpoints:

* Intracranial OR in participants with remaining non-irradiated brain metastases, as assessed by RANO-BM criteria.
* Local control rate in participants with irradiated brain metastases at 1 year, as assessed by RANO-BM criteria.
* Distant brain failure rate, the rate of new brain metastasis at a site different from the original brain metastases at 1 year, as assessed by RANO-BM criteria.
* Intracranial disease contro (CR + PR + SD) in participants with remaining non-irradiated brain metastases, as assessed by RANO-BM.

  * Intracranial clinical benefit (CR + PR + .6 months SD) in participants with remaining nonirradiated brain metastases, as assessed by RANO-BM.
  * Intracranial duration of response (DOR) in participants with remaining non-irradiated brain metastases, as assessed by the RANO-BM.
  * Time to response (TTR) in participants with remaining non-irradiated brain metastases, as assessed by the RANO-BM.
  * Safety and tolerability, as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.
  * Symptomatic radiation necrosis rate defined as the rate of clinical symptomatology requiring steroid administration and/or operative intervention concomitant with advanced and routine brain imaging findings consistent with radiation necrosis.
  * Extracranial OR, as assessed by the RECIST 1.1 and iRECIST.
  * Extracranial PFS, as assessed by the RECIST 1.1 and iRECIST.
  * Bi-compartmental PFS, as assessed by RECIST 1.1 and iRECIST for extracranial disease and RANO-BM for intracranial disease.
  * Overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants .18 years of age on the day of signing informed consent withhistologically confirmed diagnosis of RCC, irrespective of histologic will be enrolled in this study. Because no dosing or adverse event data are currently available on the use of lenvatinib in combination with pembrolizumab in patients <18 years of age, children are excluded from this study.
2. Criteria for brain metastasis:

   1. Has at least 1 measurable brain metastasis with no prior history of SRT: Presence of at least 1 independently verified, non-irradiated, measurable brain metastasis, defined as at least 5 mm AND twice the MRI slice thickness, but less than or equal to 3 cm, that can be accurately assessed at baseline and suitable for accurate repeated measurements.
   2. Has at least 1 measurable brain metastasis with prior history of SRT to other brain metastases: A history of SRT for brain metastases is allowed up to 1 week before study treatment provided that neurologic sequelae are resolved. If the patient will be enrolled to the study immediately after SRS it is encouraged to have 1-5 measurable untreated measurable lesion(s) remain, defined as at least 5 mm AND twice the MRI slice thickness, but less than or equal to 3 cm.
   3. Has no measurable brain metastasis with prior SRT: A history of immediate prior SRT for brain metastases is allowed up to 1 week before study treatment provided that neurologic sequelae are resolved.
   4. If the patient had prior SRT, progression in irradiated lesion must have occurred at least 1 month after the end of radiation therapy for the irradiated lesion to be counted as measurable.
   5. Patients can have asymptomatic (no neurologic signs or symptoms, not requiring immediate local intervention [surgery or radiosurgery] or systemic >10 mg prednisone or equivalent per day glucocorticoid therapy [within 10 days prior to study treatment initiation]) OR minimally symptomatic brain metastases (requiring .10 mg prednisone or equivalent per day and not requiring immediate surgical or radiation therapy in the opinion of the treating investigator and a radiation therapy or neurosurgical consultant).
3. Patients with brain metastasis that have not received prior systemic therapy may be eligible to enroll in this study.
4. Male participants: A male participant must agree to use a contraception as detailed in Appendix 10 of this protocol during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.
5. Female participants: A female participant is eligible to participate if she is not pregnant (see Appendix 10), not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 10 OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 10 during the treatment period and for at least 120 days after the last dose of study treatment.
6. Participants must have progressed on any prior line of treatment with an anti-PD-1/L1 mAb administered either as monotherapy or in combination with other checkpoint inhibitors or other therapies. PD-1 treatment progression is defined by meeting all of the following criteria:

   1. Has received at least 2 doses of an approved anti-PD-1/L1 mAb.
   2. Has demonstrated disease progression after anti-PD-1/L1 as defined by RECIST v1.1. The initial evidence of PD is to be confirmed by a second assessment no less than 4 weeks from the date of the first documented disease progression, in the absence of rapid clinical progression.
   3. Any number of prior treatments including anti-PD-1/L1 mAb are allowed. Anti-PD-1/L1 mAb does not have to be the most recent therapy.
7. Participants who have AEs due to previous anticancer therapies must have recovered to .Grade 1 or baseline. Participants with endocrine-related AEs who are adequately treated with hormone replacement or participants who have .Grade 2 neuropathy are eligible.
8. The participant has ability to understand and the willingness to sign a written informed consent.
9. Extracranial disease is not required and if present, it can be measurable or non-measurable (RECIST v1.1-Appendix 2).
10. Archival tumor tissue sample or newly obtained [core, incisional or excisional] biopsy of a tumor lesion not previously irradiated has been provided. FFPE tissue blocks are preferred to slides.

    Newly obtained biopsies are preferred to archived tissue.
11. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 (Appendix 4). Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
12. Has a life expectancy .12 weeks.
13. Have adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP .150/90 mm Hg with no change in antihypertensive medications within 1 week prior to study treatment.
14. Criteria for known Hepatitis B and C positive subjects

    Hepatitis B and C screening tests are not required unless:
    * Known history of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
    * As mandated by local health authority

    Hepatitis B positive subjects

    . Participants who are HBsAg positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization. . Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention.

    Participants with history of HCV infection are eligible if HCV viral load is undetectable at screening.

    • Participants must have completed curative anti-viral therapy at least 4 weeks prior to study enrollment.
15. Have adequate organ function as defined in the following table (Table 1). Specimens must be collected within 10 days prior to the start of study intervention.

Table 1 Adequate Organ Function Laboratory Values System Laboratory Value Hematological Absolute neutrophil count (ANC) .1500/ƒÊL Platelets .100 000/ƒÊL Hemoglobin .9.0 g/dL or .5.6 mmol/La Renal Creatinine OR .1.5 ~ ULN OR Measured or calculatedb creatinine clearance (GFR can also be used in place of creatinine or CrCl)

* 30 mL/min for participant with creatinine levels >1.5 ~ institutional ULN Hepatic Total bilirubin .1.5 ~ULN OR direct bilirubin .ULN for participants with total bilirubin levels >1.5 ~ ULN AST (SGOT) and ALT (SGPT) .2.5 ~ ULN (.5 ~ ULN for participants with liver metastases) Coagulation International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT)
* 1.5 ~ ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants a Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks. b Creatinine clearance (CrCl) should be calculated per institutional standard. Note: This table includes eligibility-defining laboratory value requirements for treatment; laboratory value requirements should be adapted according to local regulations and guidelines for the administration of specific chemotherapies.

Exclusion Criteria:

1. Has symptomatic brain metastasis requiring immediate procedure (surgery, radiation treatment), or corticosteroids in dosing exceeding 10 mg daily of prednisone equivalent.
2. Has received whole brain radiation treatment previously
3. Has overt hemorrhagic brain metastasis
4. Has received prior therapy with lenvatinib
5. Has clinical or radiographic evidence of leptomeningeal disease
6. Has had major surgery within 3 weeks prior to first dose of study interventions. Note: Adequate wound healing after major surgery must be assessed clinically, independent of time elapsed for eligibility. Patients must have adequately recovered from major surgery and has no ongoing surgical complications.
7. Has prior history of .Grade 3 toxicity attributed to immune checkpoint inhibitor treatment.
8. Has severe hypersensitivity (.Grade 3) to pembrolizumab and/or any of its excipients.
9. Patients must have recovered from all radiation-related toxicities, not require corticosteroids in dosing exceeding 10 mg daily of prednisone equivalent, and not have had radiation pneumonitis.
10. Active hemoptysis (bright red blood of at least 0.5 teaspoon) within 3 weeks prior to the first dose of study drug.
11. Has a history of (non-infectious, non-radiation-induced) pneumonitis not responsive to steroids or has current pneumonitis/interstitial lung disease. Patients will also be excluded if there are respiratory issues including active infection or require supplemental oxygen for activities of daily living.
12. Has preexisting .Grade 3 gastrointestinal or non-gastrointestinal fistula.
13. Gastrointestinal malabsorption or any other condition that might affect the absorption of lenvatinib
14. Has urine protein .1 g/24 hours. Note: Participants with proteinuria .2+ (.100 mg/dL) on urine dipstick testing (urinalysis) will undergo 24-hour urine collection for quantitative assessment of proteinuria.
15. Has a left ventricular ejection fraction (LVEF) below or equal to the institutional (or local laboratory) normal range, as determined by multigated acquisition (MUGA) or echocardiogram (ECHO).
16. Prolongation of the corrected QT interval by Fridericia formula (QTcF) interval to >480 ms.
17. Has clinically significant cardiovascular disease within 12 months from first dose of study intervention, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular accident, or cardiac arrhythmia associated with hemodynamic instability (Appendix 11). Note: Medically controlled arrhythmia would be permitted.
18. Contraindications to MRI (implanted metal device or foreign bodies) or MRI contrast (insufficient renal function or allergy).
19. Has a condition requiring systemic treatment with either corticosteroids (>10 mg daily) prednisone equivalent.
20. Has active autoimmune disease that has required systemic treatment in the past 3 months or a documented history of clinical severe autoimmune disease, or a syndrome that requires chronic systemic steroids or immunosuppressive agents. Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency with prednisone < 10 mg or the equivalent, etc.) is not considered a form of systemic treatment. Subjects with thyroid disease or vitiligo will not be excluded from the study.
21. Has an active infection requiring systemic therapy.
22. Has a known history of human immunodeficiency virus.
23. Has a known history of HBV (defined as hepatitis B surface antigen reactive) or known active HCV (defined as hepatitis C virus RNA [qualitative] is detected) infection.
24. Unable to swallow and retain oral medications.
25. A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation (Appendix 10). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
26. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
27. Has received prior systemic anti-cancer therapy including investigational agents within 2 weeks or 5 half-lives, whichever is shorter, prior to study treatment initiation.
28. Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
29. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
30. Known additional malignancy that is progressing or has required active treatment within the past 2 years except for except for in situ carcinoma of any site, adequately treated (without recurrence post-resection or post- radiotherapy) carcinoma of the cervix or basal or squamous cell carcinomas of the skin, or active non-threatening second malignancy that would not, in the investigator's opinion, potentially interfere with the patient's ability to participate and/or complete this trial. Examples include but not limited to urothelial cancer grade Ta or T1, adenocarcinoma of the prostate treated by active surveillance.
31. Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
32. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
33. Has had an allogenic tissue/solid organ transplant.
34. Has bleeding or thrombotic disorder(s) or uses anticoagulants such as warfarin or similar agents requiring therapeutic INR monitoring. Treatment with low molecular weight heparin is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-04 (Actual); Primary Completion 2025-08-07 (Actual); Study Completion 2025-08-07 (Actual)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jonasch, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org